CLINICAL TRIAL: NCT00069823
Title: The Study of Acid Reflux in Asthma
Brief Title: Study of Acid Reflux in Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: American Lung Association Asthma Clinical Research Centers (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Robert Wise, Professor, Johns Hopkins Bloomberg School of Public Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 157; U01HL072968 (NIH)
Record Dates: First submitted 2003-10-01; First posted 2003-10-03 (Estimated); Results first posted 2012-10-19 (Estimated); Last update posted 2012-12-19 (Estimated); Status verified 2012-12

CONDITIONS: Asthma; Lung Diseases; Lung Diseases, Obstructive
MeSH Terms: conditions — Asthma; Lung Diseases; Lung Diseases, Obstructive | interventions — Esomeprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Esomeprazole (Experimental): Proton pump inhibitor of gastric acid
  Interventions: Drug: Esomeprazole
- Placebo for esomeprazoe (Placebo Comparator): Placebo
  Interventions: Drug: Placebo proton pump inhibitor

INTERVENTIONS:
Drug: Esomeprazole — Proton pump inhibitor 40 mg orally twice daily
  Other Names: Nexium
  Arms: Esomeprazole
Drug: Placebo proton pump inhibitor — Placebo proton pump inhibitor
  Arms: Placebo for esomeprazoe

SUMMARY:
The purpose of this study is to determine if subjects with symptomatic asthma who are assigned to treatment with a proton pump inhibitor (PPI) drug such as Nexium have fewer asthma attacks than similar subjects assigned to placebo treatment.

DETAILED DESCRIPTION:
BACKGROUND:

Gastroesophageal reflux (GERD) is frequent in asthmatics with poor asthma control, often occurs without symptoms, and can induce bronchoconstriction. Poorly controlled asthmatics are often treated for GERD with drugs that suppress gastric acid, but this treatment is expensive and the benefit of such treatment is not established. Proton pump inhibitors are a relatively new class of medications that provide highly effective treatment for GERD and associated problems. This success has led many doctors to begin PPI treatment in their asthma patients in an attempt to achieve better asthma control.

DESIGN NARRATIVE:

The randomized, placebo-controlled trial will enroll 400 asthmatics, ages 18 or older, who have poor asthma control on inhaled steroids, defined on the basis of excessive bronchodilator use, nocturnal awakenings, or frequent exacerbations. Participants will be randomly assigned to treatment with either a proton pump inhibitor, esomeprazole (Nexium) 40 mg twice a day, or matching placebo. The presence, severity, and temporal relationship of GERD to asthma symptoms will be documented with 24 hour ambulatory esophageal potential Hydrogen (pH) probe monitoring, but participants will be enrolled irrespective of the severity of GERD. The primary outcome measure is the proportion of participants who have exacerbations of asthma within a 6-month period defined by asthma diaries and interviews. Secondary outcome measures include asthma symptom and control scores, asthma-specific and generic health-related quality of life, GERD symptoms, health care use, pulmonary function, and airways reactivity. Pre-specified subgroup analyses will be conducted to determine if there are clinical or demographic characteristics that predict benefit from treatment of GERD in asthma.

ELIGIBILITY:
Inclusion Criteria:

* The general goal of patient selection is to enroll patients for whom asthma physicians might prescribe GERD treatment, but where there is uncertainty whether it might be effective.
* Age 18 or older
* Physician diagnosed asthma
* If amount of air expired in the first second during a forced expiratory maneuver (FEV1) is greater than or equal to 70% predicted normal pre-bronchodilator: demonstrate methacholine 20% from post-diluent baseline (PC20). PC20 less than 16 mg/ml during Visit 1
* If FEV1 less than 70% and greater than or equal to 50% predicted normal pre-bronchodilator: demonstrate 12% reversibility during Visit 1 or within past 12 months
* Currently on stable dose of daily inhaled steroids for asthma control, i.e., inhaled corticosteroid equivalent to 400 ug/day of fluticasone44 or greater for 8 weeks or longer
* Poor asthma control: Either of the following; a score of 1.5 or greater on the Juniper Asthma Control Questionnaire; two or more episodes of asthma symptoms in the past 12 months with each episode requiring at least one of the following: an emergency department visit, unscheduled physician visit, prednisone course, hospitalization
* Non-smoker for 6 months or longer
* Less than 10 pack/year smoking history

Exclusion Criteria:

* Surgery: Previous anti-reflux or peptic ulcer surgery
* Pulmonary function: FEV1 less than 50% predicted normal pre-bronchodilator
* GERD Symptoms: Severe reflux constituting a clinical indication for treatment with a PPI or H2 blocker, typically two or more episodes per week of heartburn requiring antacids
* Other major chronic illnesses; conditions which in the judgment of the Study Physician would interfere with participation in the study, e.g., non-skin cancer, endocrine disease, coronary artery disease, congestive heart failure, stroke, severe hypertension, Type 1 insulin dependent diabetes mellitus, renal failure, liver disorders, immunodeficiency states, major neuropsychiatric disorder
* Medication use: Anti-reflux medication (proton pump inhibitors or H2 blockers) within 1 month Theophylline, azoles, iron, anti-coagulants, insulin (for Type I diabetes), digitalis, any investigative drugs within 1 month
* Drug allergy: Previous adverse effects from proton pump inhibitors or methacholine challenge
* Females of childbearing potential: Pregnant or lactating, unwilling to practice an adequate birth control method (abstinence, combination barrier and spermicide, or hormonal)
* Inability or unwillingness to provide consent
* Inability to perform baseline measurements
* Completion of less than 10 of the last 14 days of screening period diary entry
* Inability to be contacted by telephone
* Intention to move out of the area within 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 403 (Actual)
Dates: Start 2003-09; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Wise, Principal Investigator — Johns Hopkins University School of Public Health
Locations (20):
- United States (20):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California, San Diego, San Diego, California
  - National Jewish Medical and Research Center, Denver, Colorado
  - Nemours Childrens Clinic, Jacksonville, Florida
  - University of Miami, Miami, Florida
  - Emory University, Atlanta, Georgia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Indiana University ACRC, Indianapolis, Indiana
  - LSUHSC Pulmonary Critical Care, New Orleans, Louisiana
  - University of Minnesota, Minneapolis, Minnesota
  - Univ of MO Kansas City School of Medicine, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - North Shore-LIJ Medical Center, New Hyde Park, New York
  - NYU School of Medicine, New York, New York
  - New York Medical College, Valhalla, New York
  - Duke University, Durham, North Carolina
  - Ohio State University, Columbus, Ohio
  - Thomas Jefferson Hospital Pulmonary Lab, Philadelphia, Pennsylvania
  - Baylor College of Medicine, Houston, Texas
  - Northern New England Consortium, Colchester, Vermont

REFERENCES:
- [Derived] Kaminsky DA, He J, Henderson R, Dixon AE, Irvin CG, Mastronarde J, Smith LJ, Sugar EA, Wise RA, Holbrook JT. Bronchodilator response does not associate with asthma control or symptom burden among patients with poorly controlled asthma. Respir Med. 2023 Nov;218:107375. doi: 10.1016/j.rmed.2023.107375. Epub 2023 Aug 1. PMID 37536444
- [Derived] Bime C, Wei CY, Holbrook JT, Sockrider MM, Revicki DA, Wise RA. Asthma symptom utility index: reliability, validity, responsiveness, and the minimal important difference in adult asthmatic patients. J Allergy Clin Immunol. 2012 Nov;130(5):1078-84. doi: 10.1016/j.jaci.2012.07.058. Epub 2012 Sep 29. PMID 23026499
- [Derived] Bime C, Wei CY, Holbrook J, Smith LJ, Wise RA. Association of dietary soy genistein intake with lung function and asthma control: a post-hoc analysis of patients enrolled in a prospective multicentre clinical trial. Prim Care Respir J. 2012 Dec;21(4):398-404. doi: 10.4104/pcrj.2012.00073. PMID 22885561
- [Derived] DiMango E, Holbrook JT, Simpson E, Reibman J, Richter J, Narula S, Prusakowski N, Mastronarde JG, Wise RA; American Lung Association Asthma Clinical Research Centers. Effects of asymptomatic proximal and distal gastroesophageal reflux on asthma severity. Am J Respir Crit Care Med. 2009 Nov 1;180(9):809-16. doi: 10.1164/rccm.200904-0625OC. Epub 2009 Aug 6. PMID 19661245
- [Derived] American Lung Association Asthma Clinical Research Centers; Mastronarde JG, Anthonisen NR, Castro M, Holbrook JT, Leone FT, Teague WG, Wise RA. Efficacy of esomeprazole for treatment of poorly controlled asthma. N Engl J Med. 2009 Apr 9;360(15):1487-99. doi: 10.1056/NEJMoa0806290. PMID 19357404

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The planned enrollment was for 400 participants, 403 participants actually were enrolled and randomized in the trial. It is not uncommon for clinical trials not to exactly meet the sample size stated in the protocol.
Groups:
- Placebo: 40 mg of placebo twice daily
- Esomeprazole: 40 mg of esomeprazole twice daily
Period: Overall Study
Arm/Group | Placebo | Esomeprazole
Started | 199 (The design was for 200 participants per group, the study did not exactly meet the design.) | 203 (The design was for 200 participants per group, the study did not exactly meet the design.)
Completed | 193 | 200
Not Completed | 6 | 3
Not completed — Did not have follow-up diary cards | 6 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Esomeprazole | Total
Number analyzed (Participants) | 199 | 203 | 402
Age Continuous [Mean (Standard Deviation); unit: years] | 42 (13) | 42 (13) | 42 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 143 | 130 | 273
  Male | 56 | 73 | 129
Race/Ethnicity, Customized [Number; unit: participants] — Race or ethnic group was self-reported.
  participants
    White | 103 | 102 | 205
    Black | 73 | 79 | 152
    Hispanic | 17 | 18 | 35
    Other | 6 | 4 | 10
Asthma medication use [Number; unit: participants]
  Inhaled corticosteroids | 50 | 44 | 94
  Combination of fluticasone and salmeterol | 149 | 159 | 308
Body-mass index >=30 [Number; unit: participants] — The body-mass index is the weight in kilograms divided by the square of the height in meters.
  participants
    BMI >=30 | 107 | 102 | 209
    BMI <30 | 92 | 101 | 193
Conditions other than asthma [Number; unit: participants] — These conditions were self-reported.
  participants
    Gastroesophageal reflux disease | 38 | 21 | 59
    No GER reported | 161 | 182 | 343
Former smoker [Number; unit: participants]
  Former Smoker | 40 | 31 | 71
  Never smoked | 159 | 172 | 331
Health Care Visits [Number; unit: participants] — Unscheduled health care visit for asthma in previous year
  participants
    Health care visit for asthma exacerbation | 126 | 109 | 235
    No visit | 73 | 94 | 167
Pulmonary function [Number; unit: participants]
  Participants with 20% post-diluent measurement | 92 | 83 | 175
  20% from post-diluent contraindicated | 102 | 117 | 219
  Missing | 5 | 3 | 8
potential Hydrogen (pH) monitoring [Number; unit: participants] — Results of ambulatory measure of esophageal potential Hydrogen (pH) for 16 to 24 hours. Test were considered positive if pH was less than 4 for more than 5.8% of the total tiem, 8.2% of upright time, or 3.5% of supine time.
  participants
    Positive result | 62 | 61 | 123
    Negative result | 89 | 92 | 181
    Missing result | 48 | 50 | 98
%Predicted amount of air expired in the first second during a forced expiration pre broncho-dilator [Mean (Standard Deviation); unit: Percent] — Percent of the predicted value for the amount of air expired in the first second during a forced expiratory maneuver (FEV1) based on gender, age and ethnicity that the measured value is.
  Percent | 78 (15) | 76 (16) | 77 (16)
Age of onset of asthma [Mean (Standard Deviation); unit: years] | 17 (17) | 17 (16) | 17 (16)
Age of participants [Mean (Standard Deviation); unit: years]
  at randomization | 42 (13) | 42 (13) | 42 (13)
  at onset of asthma | 17 (17) | 17 (16) | 17 (16)
Asthma scores [Mean (Standard Deviation); unit: score] — Asthma Control Score (ACS)ranges from 0 to 6, lower scores indicating better asthma control and 0.5 as the minimal clinically important difference; Asthma Symptom Utility Index (ASUI) score ranges from 0 to 1, higher scores indicating less severe asthma; Mini-Asthma Quality of Life Questionnaire (mini-AQLQ) score range from 1 to 7, higher scores indicating better quality of life and 0.5 as the minimal clinically important difference.
  score
    ACQ | 1.9 (0.8) | 1.8 (0.8) | 1.8 (0.8)
    ASUI | 0.74 (0.18) | 0.76 (0.15) | 0.75 (0.15)
    mini asthma quality of life questionnaire | 4.7 (1.2) | 4.7 (1.2) | 4.7 (1.2)
Percent change in FEV1 after bronchodilator [Mean (Standard Deviation); unit: Percent change] — The percent difference in FEV1 before and after using a bronchodilator (albuterol) divided by the value before bronchodilation.
  Percent change | 10 (10) | 11 (16) | 11 (13)

OUTCOME MEASURES:

1. Secondary Outcome: Exacerbation Components: >=30% Drop in Peak Expiratory Flow on 2 Consecutive Days
Time Frame: Baseline to 24 Weeks
Measure: Number; unit: events per person-year
Arm/Group | Placebo | Esomeprazole
Number analyzed (Participants) | 193 | 200
events per person-year | 1.7 | 2.1
Statistical Analysis 1: Comparison: Placebo vs Esomeprazole; Rates were compared with incidence-rate ratios (IRR). The IRR and P values were estimated with the use of negative binomial regression models with robust variance estimates; Test type: Superiority or Other; p = 0.35, Negative binomial regression — P values are for the treatment effect of esomeprazole as compared with placebo; Incidence-Rate Ratio = 1.2, 95% CI 2-sided [0.8 to 2.0]

2. Secondary Outcome: Exacerbation Components: Urgent Care Visit
Time Frame: Measured at Month 6
Measure: Number; unit: events per person-year
Arm/Group | Placebo | Esomeprazole
Number analyzed (Participants) | 193 | 200
events per person-year | 0.6 | 0.5
Statistical Analysis 1: Comparison: Placebo vs Esomeprazole; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.79, Negative binomial regression — P values are for the treatment effect of esomeprazole as compared with placebo; Incidence-Rate Ratio = 0.9, 95% CI 2-sided [0.6 to 1.5]

3. Primary Outcome: Episodes of Poor Asthma Control (EPAC) From Diary Cards, According to Definition That Did Not Include Use of Beta-agonists as a Criterion
Description: Episodes of poor asthma control was defined as any one of the following: 2 consecutive days with a drop in peak flow >=30% of baseline; urgent care for asthma; or new use of oral corticosteroids for asthma
Time Frame: Baseline to 24 Weeks
Measure: Number; unit: events per person year
Arm/Group | Placebo | Esomeprazole
Number analyzed (Participants) | 193 | 200
events per person year | 2.3 | 2.5
Statistical Analysis 1: Comparison: Placebo vs Esomeprazole; The rates of EPACs were compared using incidence-rate ratios (IRR). IRR and P value were estimated with the use of negative binomial regression models with robust variance estimates; Test type: Superiority or Other; p = 0.66, Negative binomial regression — P values are for the treatment effect of esomeprazole as compared with placebo; Incidence-Rate Ratio = 1.1, 95% CI 2-sided [0.8 to 1.5]

4. Secondary Outcome: Exacerbation Components: New Use of Oral Corticosteroids
Time Frame: Baseline to 24 Weeks
Measure: Number; unit: events per person year
Arm/Group | Placebo | Esomeprazole
Number analyzed (Participants) | 193 | 200
events per person year | 0.6 | 0.5
Statistical Analysis 1: Comparison: Placebo vs Esomeprazole; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.62, Negative binomial regression — P values are for the treatment effect of esomeprazole as compared with placebo; Incidence-Rate Ratio = 0.9, 95% CI 2-sided [0.6 to 1.3]

5. Secondary Outcome: Asthma Episodes, According to Definition That Included Increased Use of Beta-agonists
Time Frame: Baseline to 24 Weeks
Measure: Number; unit: events per person-year
Arm/Group | Placebo | Esomeprazole
Number analyzed (Participants) | 193 | 200
events per person-year | 4.4 | 4.3
Statistical Analysis 1: Comparison: Placebo vs Esomeprazole; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.87, Negative binomial regression — P values are for the treatment effect of esomeprazole as compared with placebo; Incidence-Rate Ratio = 1.0, 95% CI 2-sided [0.8 to 1.3]

6. Secondary Outcome: Use of Rescue Medications
Description: Increase in the use of rescue meds by 4 or more uses on a particular day above the average uses during the run-in period.
Time Frame: Baseline to 24 Weeks
Measure: Number; unit: events per person-year
Arm/Group | Placebo | Esomeprazole
Number analyzed (Participants) | 193 | 200
events per person-year | 3.0 | 2.8
Statistical Analysis 1: Comparison: Placebo vs Esomeprazole; Incidence-rate ratios and P values were estimated with the use of negative binomial regression models with robust variance estimates; Test type: Superiority or Other; p = 0.62, Negative binomial regression — P values are for the treatment effect of esomeprazole as compared with placebo; Incidence-Rate Ratio = 0.9, 95% CI [0.7 to 1.3]

7. Secondary Outcome: Night Awakening
Description: Rate of awakening at night because of asthma symptoms
Time Frame: Baseline to 24 Weeks
Measure: Number; unit: events per person-year
Arm/Group | Placebo | Esomeprazole
Number analyzed (Participants) | 193 | 200
events per person-year | 30 | 28
Statistical Analysis 1: Comparison: Placebo vs Esomeprazole; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.70, Negative binomial regression — P values are for the treatment effect of esomeprazole as compared with placebo; Incidence-Rate Ratio = 0.9, 95% CI 2-sided [0.6 to 1.4]

8. Secondary Outcome: Pulmonary Function: Change in Prebronchodilator FEV1
Description: Mean change in pre-bronchodilator FEV1 - forced expiratory volume in 1 second; a measure of pulmonary function. The treatment effect is the difference in the mean change in between the groups.
Time Frame: Baseline to 24 Weeks
Population: The analyses are based on data from 191 participants in the placebo group and 201 in the esomeprazole group, with the following exception: 41 participants in the placebo group and 37 in the esomeprazole group for measurement of 20% post-diluent baseline (PC20).
Measure: Mean (95% Confidence Interval); unit: liters
Arm/Group | Placebo | Esomeprazole
Number analyzed (Participants) | 191 | 201
liters | -0.02 [-0.06 to 0.01] | 0.00 [-0.04 to 0.04]
Statistical Analysis 1: Comparison: Placebo vs Esomeprazole; The treatment effect is the mean change in the Esomeprazole group - mean change in placebo group; Test type: Superiority or Other; p = 0.36, Regression, Linear — P values were calculated with the use of linear regression; Mean Difference (Net) = 0.03, 95% CI 2-sided [-0.03 to 0.08], Standard Error of Mean 0.03 — Treatment effect is the difference in mean change in the esomeprazole group minus the mean change in the placebo group, e.g. 0.00 - (-0.02) = -0.03 (rounding)

9. Secondary Outcome: Pulmonary Function: Change in Prebronchodilator Forced Vital Capacity
Description: Pulmonary function measured by mean change in Prebronchodilator forced vital capacity from baseline to 24 weeks
Time Frame: Baseline to 24 Weeks
Measure: Mean (95% Confidence Interval); unit: liters
Arm/Group | Placebo | Esomeprazole
Number analyzed (Participants) | 191 | 201
liters | -0.03 [-0.06 to 0.01] | 0.00 [-0.04 to 0.05]
Statistical Analysis 1: Comparison: Placebo vs Esomeprazole; Test type: Superiority or Other; p = 0.30, Regression, Linear; Mean Difference (Final Values) = 0.03, 95% CI 2-sided [-0.03 to 0.09], Standard Error of Mean 0.03 — Treatment effect is the difference in mean change in the esomeprazole group minus the mean change in the placebo group

10. Secondary Outcome: Pulmonary Function: Change in Peak Flow Rate
Description: Mean change from baseline to 24 weeks in the peak flow rate - how forceful patient can blow out air
Time Frame: Baseline to 24 Weeks
Measure: Mean (95% Confidence Interval); unit: liters/min
Arm/Group | Placebo | Esomeprazole
Number analyzed (Participants) | 191 | 201
liters/min | 3.2 [-3.5 to 9.9] | 9.2 [1.8 to 16.6]
Statistical Analysis 1: Comparison: Placebo vs Esomeprazole; Test type: Superiority or Other; p = 0.24, Regression, Linear; Mean Difference (Final Values) = 6.0, 95% CI 2-sided [-4.0 to 16.0], Standard Error of Mean 5.1 — Treatment effect is the difference in mean change in the esomeprazole group minus the mean change in the placebo group

11. Secondary Outcome: Pulmonary Function: Change in PC20
Description: Mean Change in the dose of methacholine that results in a 20% drop in FEV1
Time Frame: Baseline to 24 Weeks
Measure: Mean (95% Confidence Interval); unit: mg/ml
Arm/Group | Placebo | Esomeprazole
Number analyzed (Participants) | 41 | 37
mg/ml | 1.5 [0.2 to 2.9] | 0.3 [-1.4 to 0.9]
Statistical Analysis 1: Comparison: Placebo vs Esomeprazole; Test type: Superiority or Other; p = 0.04, Regression, Linear; Treatment Effect = -1.8, 95% CI [-3.6 to -0.1]

12. Secondary Outcome: Change in Juniper Asthma Control Score(JACQ)
Description: Mean change. Scores on the JACQ range from 0 to 6, with lower scores indicating better asthma control and 0.5 as the minimal clinically important difference.
Time Frame: Baseline to 24 Weeks
Measure: Mean (95% Confidence Interval); unit: score
Arm/Group | Placebo | Esomeprazole
Number analyzed (Participants) | 191 | 201
score | -0.3 [-0.4 to -0.2] | -0.2 [-0.3 to -0.1]
Statistical Analysis 1: Comparison: Placebo vs Esomeprazole; Test type: Superiority or Other; p = 0.11, Regression, Linear; Treatment Effect = 0.1, 95% CI 2-sided [0.0 to 0.2], Standard Error of Mean 0.1 — Treatment effect is the difference in mean change in the esomeprazole group minus the mean change in the placebo group

13. Secondary Outcome: Change in Asthma Symptom Utility Index (ASUI)
Description: Mean change. Scores on the ASUI range from 0 to 1, with higher scores indicating less severe asthma.
Time Frame: Baseline to 24 Weeks
Measure: Mean (95% Confidence Interval); unit: score
Arm/Group | Placebo | Esomeprazole
Number analyzed (Participants) | 191 | 201
score | 0.05 [0.03 to 0.07] | 0.02 [0.01 to 0.04]
Statistical Analysis 1: Comparison: Placebo vs Esomeprazole; Test type: Superiority or Other; p = 0.11, Regression, Linear; Mean Difference (Final Values) = -0.02, 95% CI 2-sided [-0.05 to -0.02], Standard Error of Mean 0.01 — Treatment effect is the difference in mean change in the esomeprazole group minus the mean change in the placebo group

14. Secondary Outcome: Change in the Mini-Asthma Quality of Life Questionnaire (Mini-AQLQ)
Description: Mean change. Scores on the Mini-Asthma Quality of Life Questionnaire (mini-AQLQ)range from 1 to 7, with higher scores indicating better quality of life and 0.5 as the minimal clinically important difference.
Time Frame: Baseline to 24 Weeks
Measure: Mean (95% Confidence Interval); unit: score
Arm/Group | Placebo | Esomeprazole
Number analyzed (Participants) | 191 | 201
score | 0.3 [0.2 to 0.4] | 0.3 [0.2 to 0.4]
Statistical Analysis 1: Comparison: Placebo vs Esomeprazole; Test type: Superiority or Other; p = 0.33, Regression, Linear; Mean Difference (Net) = -0.1, 95% CI 2-sided [-0.2 to 0.1], Standard Error of Mean 0.1 — Treatment effect is the difference in mean change in the esomeprazole group minus the mean change in the placebo group

15. Secondary Outcome: Change in Medical Outcomes Study Short-Form 36 Score Quality of Life Score: Physical Component
Description: Mean change. Scores on the Medical Outcomes Study Short-Form 36 range from 1 to 100, with higher scores indicating better quality of life and 5 as the minimal clinically important difference.
Time Frame: Baseline to 24 Weeks
Measure: Mean (95% Confidence Interval); unit: score
Arm/Group | Placebo | Esomeprazole
Number analyzed (Participants) | 191 | 201
score | 2.0 [1.1 to 2.9] | 1.1 [0.3 to 1.9]
Statistical Analysis 1: Comparison: Placebo vs Esomeprazole; Test type: Superiority or Other; p = 0.16, Regression, Linear; Mean Difference (Net) = -0.9, 95% CI 2-sided [-2.0 to 0.4], Standard Error of Mean 0.6 — Treatment effect is the difference in mean change in the esomeprazole group minus the mean change in the placebo group

16. Secondary Outcome: Change in Medical Outcomes Study Short-Form 36 Quality of Life Score: Mental Component
Description: as for outcome 15
Time Frame: Baseline to 24 Weeks
Measure: Mean (95% Confidence Interval); unit: score
Arm/Group | Placebo | Esomeprazole
Number analyzed (Participants) | 191 | 201
score | 0.0 [-1.8 to 1.1] | 0.4 [-0.5 to 1.4]
Statistical Analysis 1: Comparison: Placebo vs Esomeprazole; Test type: Superiority or Other; p = 0.56, Regression, Linear; Mean Difference (Net) = 0.5, 95% CI 2-sided [-1.1 to 2.2], Standard Error of Mean 0.78 — Treatment effect is the difference in mean change in the esomeprazole group minus the mean change in the placebo group

17. Secondary Outcome: Change in Gastric Symptoms: Gastroesophageal Reflux Disease Symptom Assessment Scale Score
Description: Mean change. The Gastroesophageal Reflux Disease Symptom Assessment Scale score ranges from 0 to 3, with lower numbers indicating less distress.
Time Frame: Baseline to 24 Weeks
Measure: Mean (95% Confidence Interval); unit: score
Arm/Group | Placebo | Esomeprazole
Number analyzed (Participants) | 191 | 201
score | -0.17 [-0.21 to -0.12] | -0.16 [-0.20 to -0.11]
Statistical Analysis 1: Comparison: Placebo vs Esomeprazole; Test type: Superiority or Other; p = 0.76, Regression, Linear; Mean Difference (Net) = 0.01, 95% CI 2-sided [-0.05 to 0.07], Standard Error of Mean 0.03 — Treatment effect is the difference in mean change in the esomeprazole group minus the mean change in the placebo group

18. Secondary Outcome: Change in Number of Gastric Symptoms: No. of Symptoms
Description: Mean change
Time Frame: Baseline to 24 Weeks
Measure: Mean (95% Confidence Interval); unit: symptoms
Arm/Group | Placebo | Esomeprazole
Number analyzed (Participants) | 191 | 201
symptoms | -1.7 [-2.1 to -1.3] | -1.9 [-2.3 to -1.6]
Statistical Analysis 1: Comparison: Placebo vs Esomeprazole; Test type: Superiority or Other; p = 0.39, Regression, Linear; Mean Difference (Net) = -0.2, 95% CI 2-sided [-0.8 to 0.3], Standard Error of Mean 0.3 — Treatment effect is the difference in mean change in the esomeprazole group minus the mean change in the placebo group

ADVERSE EVENTS:
Arm/Group | Placebo | Esomeprazole
Serious Adverse Events (participants affected / at risk) | 16/199 | 10/203
Other Adverse Events (participants affected / at risk) | 0/199 | 0/203
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo (N=199) | Esomeprazole (N=203)
Asthma exacerbation requiring hospitalization (Respiratory, thoracic and mediastinal disorders) | 4/193 (4) | 3 (3)
Hospitalization or emergency department visit for surgery, trauma, or other acute illness (General disorders) | 9/193 (10) | 5 (6)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0/193 (0) | 1 (1)
Death from complications after surgery for endobronchial tumor (Respiratory, thoracic and mediastinal disorders) | 0/193 (0) | 1 (1)
Hospitalization for possible cardiac ischemia (Cardiac disorders) | 2/193 (2) | 0 (0)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1/143 (1) | 0/130 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No